CLINICAL TRIAL: NCT05143424
Title: Phase 1 Drug-drug Interaction of Cannabidiol and Morphine in Recreational Opioid Users
Brief Title: Evaluation of the Interactions of Cannabidiol (CBD) With Morphine
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: NIDA-CBD-Phase1a-002
Record Dates: First submitted 2021-11-09; First posted 2021-12-03 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Opioid Use Disorder
Keywords: Marijuana Abuse; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorders; Central Nervous System Depressants; Psychotropic Drugs; Neurotransmitter Agents; Cannabidiol; CBD; Morphine; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Opioid-Related Disorders; Marijuana Abuse; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorders | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBD (350 mg) (Active Comparator): CBD 350 mg twice per day for 3 days
  Interventions: Drug: Morphine Sulfate
- CBD (700 mg) (Active Comparator): CBD 700 mg twice per day for 3 days
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Morphine Sulfate — Morphine sulfate 30 mg tablets as a single dose twice
  Other Names: Placebo oral capsule; Placebo

SUMMARY:
The purpose of this study is to analyze drug-drug interactions of CBD on co-administered Morphine as first step in understanding CBD-opioid interactions.

DETAILED DESCRIPTION:
This is an inpatient, single-blind, non-randomized, 1-sequence study involving healthy subjects who have used opioids for recreational use. The primary objective of the study is to establish the pharmacokinetic parameters of morphine 30 mg when administered with and without CBD 350 mg b.i.d. and CBD 700 mg b.i.d.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and provide written informed consent prior to the initiation of any protocol-specific procedures.
* Males and females 18 to 55 years of age, inclusive.
* Body mass index (BMI) ranging from 18 to 34 kg/m2, inclusive, and body weight of 56 kg and above.
* Adequate venous access as assessed by an investigator at screening.
* No clinically significant concurrent medical conditions determined by medical history, physical examination, clinical laboratory examination, vital signs, and 12-lead ECG.
* Recreational opioid use (i.e., defined as prescription opioid use for nontherapeutic purposes on at least 3 occasions within the previous year and at least once in the 12 weeks prior to screening), experienced in using opioids of approximately 30 mg morphine equivalents and not seeking treatment for Opioid Use Disorder.
* If of childbearing potential, a female study subject must agree to use 1 of the accepted contraceptive regimens from at least 30 days prior to the first administration of the study medication, during the study and for at least 30 days after the last dose of the study medication

  1. An acceptable method of contraception includes abstinence from heterosexual intercourse or intrauterine device (with or without hormones)
  2. OR agrees to use a double barrier method (e.g., condom and spermicide) during the study and for at least 30 days after the last dose of the study medication. Oral contraceptives are prohibited.
  3. If a female of non-childbearing potential, she should be surgically sterile (i.e., has undergone compete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least 1 year without menses), as confirmed by FSH level.
* A male study subject must agree to use a double barrier method (e.g., condom and spermicide) and agree to not donate sperm during the study and for at least 90 days after the last dose of the study medication.
* Agree not to ingest alcohol, drinks containing caffeine >500 mg/day (e.g., Coca Cola®, tea, coffee, etc.), or grapefruit/grapefruit juice or participate in strenuous exercise 72 hours prior to admission through the last blood draw of the study.
* Able to speak, read, and understand English sufficiently to allow completion of all study assessments.
* Must be willing and able to abide by all study requirements and restrictions.

Exclusion Criteria:

* Contact site directly for more information

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Establish the Maximum Plasma Concentration (Cmax) of morphine when administered orally with and without CBD | 3 day
  Establish the Maximum Plasma Concentration (Cmax) of morphine when administered orally with and without CBD 350 mg b.i.d. and CBD 700 mg b.i.d.
Establish the Area Under the Curve (AUC 0-t) of morphine and its 2 glucuronide conjugates when morphine is administered with and without CBD | 3 day
  Establish the Area Under the Curve (AUC 0-t) of morphine and its 2 glucuronide conjugates when morphine is administered with and without CBD 350 mg b.i.d. and CBD 700 mg b.i.d.
Establish the Area Under the Curve from zero to infinity (AUC 0-inf) of morphine and its 2 glucuronide conjugates when morphine is administered with and without CBD | 3 day
  Establish the Area Under the Curve from zero to infinity (AUC 0-inf) of morphine and its 2 glucuronide conjugates when morphine is administered with and without CBD 350 mg b.i.d. and CBD 700 mg b.i.d.

SECONDARY OUTCOMES:
Establish the Time of Maximum Plasma Concentration (Tmax) of morphine when administered orally with and without CBD | 3 day
  Establish the Time of Maximum Plasma Concentration (Tmax) of morphine when administered orally with and without CBD 350 mg b.i.d. and CBD 700 mg b.i.d.
Establish the Terminal Phase Elimination Rate Constant of morphine when administered orally with and without CBD | 3 day
  Establish the Terminal Phase Elimination Rate Constant of morphine when administered orally with and without CBD 350 mg b.i.d. and CBD 700 mg b.i.d.
Establish the Apparent Clearance of morphine when administered orally with and without CBD | 3 day
  Establish the Apparent Clearance of morphine when administered orally with and without CBD 350 mg b.i.d. and CBD 700 mg b.i.d.
Establish the Maximum Plasma Concentration (Cmax) of CBD when administered orally with morphine | 3 day
  Establish the Maximum Plasma Concentration (Cmax) of CBD 350 mg b.i.d. and CBD 700 mg b.i.d. when administered orally with morphine
Establish the Time of Maximum Plasma Concentration (Tmax) of CBD when administered orally with morphine | 3 day
  Establish the Time of Maximum Plasma Concentration (Tmax) of CBD 350 mg b.i.d. and CBD 700 mg b.i.d. when administered orally with morphine
Establish the Area Under the Curve of the dosing period of CBD when administered orally with morphine | 3 day
  Establish the Area Under the Curve of the dosing period of CBD 350 mg b.i.d. and CBD 700 mg b.i.d. when administered orally with morphine
Establish the Apparent Clearance of CBD when administered orally with morphine | 3 day
  Establish the Apparent Clearance of CBD 350 mg b.i.d. and CBD 700 mg b.i.d. when administered orally with morphine
Establish the terminal half-life of CBD when administered orally with morphine | 3 day
  Establish the terminal half-life of CBD 350 mg b.i.d. and CBD 700 mg b.i.d. when administered orally with morphine
Establish the terminal-phase elimination rate constant of CBD when administered orally with morphine | 3 day
  Establish the terminal-phase elimination rate constant of CBD 350 mg b.i.d. and CBD 700 mg b.i.d. when administered orally with morphine
Safety and Tolerability of morphine when administered orally with or without CBD by collecting vital signs and recording treatment emergent adverse events | 7 + 3/5 days
  Incidence of treatment Emergent Adverse Events using the most recent version of the Medical Dictionary of Regulatory Activities (MedDRA) preferred terms, its relationship to the treatment, and maximum severity, either reported by the subject or by clinically significant abnormal findings on:
  i. Physical examination ii. Rate of change in vital signs assessments of heart rate, sitting blood pressure, respiration rate, and temperature iii. Rate of change in ECG assessment iv. Rate of change in venous CO2 concentrations v. Rate of clinical laboratory changes

CONTACTS AND LOCATIONS:
Locations (1):
- AltaSciences, Overland Park, Kansas, United States